CLINICAL TRIAL: NCT00747825
Title: A Phase I Study Evaluating the Safety, Pharmacokinetics, Tissue Distribution, and Determination of Radiation Dosimetry for 131-I-MIP-1145
Brief Title: Phase I Safety and Dosimetry Study in Patients With Confirmed Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SZ-M101
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Metastatic Melanoma
Keywords: cancer; oncology; melanoma; tumor
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — N-(2-diethylaminoethyl)-4-(4-fluorobenzamido)-5-iodo-2-methoxybenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 131-I-MIP-1145 — IV injection between 4.0 to 6.0 mCi (148-222 MBq) of 131-I-MIP-1145

SUMMARY:
This is an open-label, single dose study for patients 18 years of age or older with confirmed metastatic melanoma. Up to 12 patients will be enrolled and all will receive an injection of approximately 4.0 to 6.0 mCi (148-222 MBq) of 131-I-MIP-1145 administered via IV injection. The study will consist of a single dosing day followed by a 7-day assessment period and 21-day follow-up period. The total duration of the study from screening to final follow-up visit is approximately 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and be willing to comply with all protocol requirements
2. Men and women 18 years of age or older
3. Female patients must meet 1 of the following criteria:

   * not be of childbearing potential as documented by medical history (e.g., tubal ligation or hysterectomy), or be post menopausal with a minimum 1 year without menses
   * Have a negative serum beta human chorionic gonadotropin (BHCG) pregnancy test within 48 hours prior to receiving the test article and agree to use a medically acceptable form of birth control, defined as abstinence or use of an intrauterine device (IUD), oral contraceptive, barrier and spermicide, or hormonal implant throughout the 28 day study period.
4. Male patients of childbearing potential must agree to use at least one of the following medically acceptable forms of birth control throughout the 28 day study period; abstinence, barrier or other acceptable, effective contraceptive method.
5. Historical diagnosis (surgical or histological) of primary melanoma with metastatic melanoma confirmed by histology and/or radiologically via MRI/CT.
6. CT/MRI representing current measurable metastatic lesion (within 6 to 12 weeks of entry; at least one lesion > 2cm in the longest dimension)

Exclusion Criteria:

1. Less than 18 years of age
2. Pregnant or breastfeeding
3. Inadequate venous access (defined as contralateral antecubital or equivalent venous access sites which are required for study drug injection and PK blood sampling, respectively)
4. Uncontrolled glaucoma or retinopathy (e.g. macular degeneration) treated in the past year
5. Cataracts or other lens opacities
6. Any ophthalmologic intervention within the last 30 days (e.g., cataract extraction, laser procedure or equivalent, anti-VEGF treatment for macular degeneration. Topical treatments including antibiotics for conjunctivitis are allowed.)
7. Patient received external beam therapy or chemotherapy within the last 30 days
8. Any history of head and neck radiotherapy
9. Karnofsky performance status is less than 60 (ECOG status > 2)
10. Serum creatinine is greater or equal to 2.0 mg/dL
11. Total bilirubin greater or equal to 1.5 times upper limit of normal
12. SGOT/AST or SGPT/ALT greater or equal to 3 times upper limit of normal (patients with metastatic liver disease are eligible if transaminase elevation is > 5 times the upper limit of normal)
13. Received an investigational compound and/or medical device within 30 days before admission into this study
14. Administered a 99mTc-labeled radioisotope < 3 days prior to imaging or < 7days prior to imaging for other diagnostic radioisotopes with half lives greater than 24 hours
15. Any known allergy or sensitivity to iodine. Iodinated X-ray contrast hypersensitivity is not an exclusion.
16. Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-injection follow-up examinations
17. Determined by the Investigator to be clinically unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

SECONDARY OUTCOMES:
To estimate radiation absorbed doses (dosimetry) to known 131-I-MIP-1145 avid lesions and to the whole body, following a single bolus (IV) injection of approximately 4.0 to 6.0 mCi (148-222 MBq) of 131-I-MIP-1145.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States